CLINICAL TRIAL: NCT01442831
Title: An Open-label Study to Evaluate the Absorption, Metabolism, and Excretion of Orally Administered [14C]-TR-701 in Healthy Adult Male Subjects
Brief Title: Evaluate the Absorption, Metabolism, And Excretion Of Orally Administered [14C] TR 701 In Healthy Adult Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trius Therapeutics LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1986-024; TR701-106 (Other: TriusRX unique Id)
Record Dates: First submitted 2011-06-06; First posted 2011-09-29 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Healthy
Keywords: metabolic profile of TR-700 in plasma urine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Human ADME (Experimental)
  Interventions: Drug: Human ADME

INTERVENTIONS:
Drug: Human ADME — Oral single dose

SUMMARY:
The purpose of this study is to describe the single dose pharmacokinetics of total radioactivity in plasma and whole blood following PO administration of [14C] TR-701 in healthy adult male subjects.

DETAILED DESCRIPTION:
This study will be an open-label, single-dose study of the absorption, metabolism, and excretion of 200 mg [14C]-TR-701 (approximately 100 μCi) administered orally following at least an 8-hour fast. Subjects will receive a single dose of 200 mg [14C] TR 701 (approximately 100 μCi) administered as an oral solution.

The dose will be administered following at least an 8-hour fast and followed by a 4-hour fast from food, not including water.

ELIGIBILITY:
Inclusion Criteria:

1. Males, between 18 and 50 years of age, inclusive.
2. Body mass index (BMI) of 20 kg/m2 to 29.9 kg/m2, inclusive.
3. In good health, determined by no clinically significant findings from medical history, physical examination (Check-in), 12-lead ECG, and vital signs.

Exclusion Criteria:

1. Significant history or clinical manifestation of any significant metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder (as determined by the Investigator and Sponsor).
2. History of an abnormal ECG that is clinically significant in the opinion of the Investigator.
3. History of hypersensitivity, intolerance, or allergy to antibiotics of the oxazolidinone class, to any ingredient of the formulation.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2010-09-09 (Actual); Primary Completion 2010-09-22 (Actual); Study Completion 2010-09-22 (Actual)

PRIMARY OUTCOMES:
To describe the single dose plasma PK of TR-700, the microbiologically active molecule | pre dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, then daily up to 312 hours post dose
  To describe the single dose pharmacokinetics (Cmax, Tmax, AUC, t 1/2, CL/F) of total radioactivity in plasma, whole blood, urine and feces following oral (PO) administration of [14C] TR 701 in healthy adult male subjects

CONTACTS AND LOCATIONS:
Overall Officials: Philippe G Prokocimer, MD, Study Chair — Trius Therapeutics
Locations (1):
- Trius Investigator Site 001, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Ong V, Flanagan S, Fang E, Dreskin HJ, Locke JB, Bartizal K, Prokocimer P. Absorption, distribution, metabolism, and excretion of the novel antibacterial prodrug tedizolid phosphate. Drug Metab Dispos. 2014 Aug;42(8):1275-84. doi: 10.1124/dmd.113.056697. Epub 2014 May 29. PMID 24875463